CLINICAL TRIAL: NCT01512238
Title: Improvement of Intentional and Unintentional Non-adherence in the Elderly. Importance of Pharmaceutical Care, Generic Substitution, Non-prescription Drugs, Herbal Medicine and Dietary Supplements
Brief Title: Improvement of Intentional and Unintentional Non-adherence in the Elderly
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: CO01
Record Dates: First submitted 2012-01-04; First posted 2012-01-19 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2013-12

CONDITIONS: Medication Adherence
Keywords: Medicine adherence; Drug substitution; Herb-drug interaction; Herbal medicine; Dietary supplements; Over-the-counter products; On-line prescription records; Personal electronic medicine profile; Intentional non-adherence; Unintentional non-adherence
MeSH Terms: conditions — Medication Adherence | interventions — Pharmaceutical Services

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pharmaceutical care
  Interventions: Other: Pharmaceutical care
- Control

INTERVENTIONS:
Other: Pharmaceutical care — Information about medicine, sideeffect, adherence
  Other Names: Pharmaceutical Services
  Groups: Pharmaceutical care

SUMMARY:
The purpose is to study if different factors influence medicine adherence in elderly people. In this study number of generic substitution and use of non-prescription drugs, herbal medicine and dietary supplement is in focus.

DETAILED DESCRIPTION:
The purpose of this study is to describe in the elderly:

1. Association between medicine adherence and number of generic substitution
2. Association between medicine adherence and use of non-prescription drugs, herbal medicine and dietary supplements and interaction between 'prescription drugs' and 'non-prescription drugs, herbal medicine and dietary supplements'
3. Intentional and unintentional non-adherence

Some of the data in the present study were originally collected as part of a major research project 'Methods for Improving Compliance with Medicine Intake' (MICMI). The study sample of 945 persons was randomly selected into three groups: two intervention groups and one control group. Interventions were pharmaceutical care and an electronic reminder system. All groups were followed for one year.

Data in the present study is from the pharmaceutical care group and the control group, and is descriptive.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Living in their own homes
* Without assistance to medicine administration
* Living in the Municipality of Aarhus, Denmark
* Long-term treatment with > 4 prescription drugs

Exclusion Criteria:

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Persons aged 65 years or older, living in their own homes without assistance to medicine administration in the Municipality of Aarhus, Denmark and who were in long-term treatment with > 4 prescription drugs at the beginning of the project
Sampling Method: Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Medicine adherence | One year

SECONDARY OUTCOMES:
Number of generic substitution | One year
Use of non-prescription drugs, herbal medicine and dietary supplements and frequency of interaction between 'prescription drugs' and 'non-prescription drugs, herbal medicine and dietary supplements' | Actually day
Intentional and unintentional non-adherence association with generic substitution and use of non-prescription drugs, herbal medicine and dietary supplements | One year

CONTACTS AND LOCATIONS:
Overall Officials: Else Marie S Damsgaard, Professor, Study Chair — Aarhus University Hospital; Ishay Barat, Ph.D., Study Chair — Horsens Hospital